CLINICAL TRIAL: NCT03680027
Title: Effects Of Walnut-Enriched Diet On Blood Lipids And Glucose Profiles In Hyperlipidemic Subjects: A Randomized-Controlled Trial: A Randomized-Controlled Trial
Brief Title: Effects Of Walnut-Enriched Diet On Blood Lipids And Glucose Profiles In Hyperlipidemic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gözde Okburan, Senior Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/13-04
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Hyperlipidemias
Keywords: Serum lipids; Hyperlipidemia; Walnut
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): In 'Control group' participants had 6 week follow-up without any intervention.
- Interventional Group (Experimental): In 'Interventional group' participants had 6 week follow-up and during that period of time, they were asked to consume 40g/day walnut. Participants in intervention group was ensured to consume all 40g of walnut every day, during their snack times for 6 weeks.
  Interventions: Dietary Supplement: Walnut-enriched Group

INTERVENTIONS:
Dietary Supplement: Walnut-enriched Group — All subjects supplemented with 40 g/day of walnuts for 6 weeks.
  Arms: Interventional Group

SUMMARY:
Walnuts have been shown to reduce serum lipids in hyperlipidemic individuals with a well-controlled feeding trials. Current study have been determined the effects of daily walnut consumption on serum lipids, fasting glucose and insulin levels in hyperlipidemic individuals.

DETAILED DESCRIPTION:
In this, randomized controlled trial, mild to moderate hyperlipidemic subjects were randomly divided into 2 groups as walnut-enriched (n=20) and control (n=17) groups for 6 weeks. All subjects adhered to a medical nutrition therapy as low-fat and low-cholesterol diet. The walnut-enriched group was supplemented with 40 g/day of walnuts added to their diets. In order to follow nutritional status of subjects, they were visited every 15 days (in total 4 times). Anthropometric measurements of the subjects were taken and were monitored at each visit during the study. Blood samples were measured at the beginning and again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemic patients who are not using any lipid lowering medications
* Non-smoker
* No alcohol consumption
* Individuals who are having ≤30kg/m2
* Individuals who do not have any allergy for nut consumption
* Female participants who are not pregnant or breastfeeding
* Individuals should not be in a weight loss programme
* Having not consumed regular nuts for the last 1 month,
* Except hypertension, they should not have other chronic diseases (such as diabetes, chronic renal failure)
* No intense exercise

Exclusion Criteria:

* Failure to meet the criteria for inclusion criteria.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction in serum lipids and fasting glucose levels | Six weeks
  In both group, participants have decreased serum total cholesterol and LDL-cholesterol.However especially walnut-enrcihed group significantly changed fasting glucose and insulin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Okburan, Principal Investigator — Eastern Mediterranean University

IPD SHARING:
Plan to Share IPD: Undecided